CLINICAL TRIAL: NCT02500017
Title: Melatonin Treatment for Night-Eating Syndrome
Acronym: MLT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting appropriate participants
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Cenk Tek, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1503015417
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Night-eating Syndrome
MeSH Terms: conditions — Night Eating Syndrome | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Experimental): A commercially available rapid-release formulation of melatonin (5 mg) capsules to be administered once a day for a total of 8 weeks
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): Matching placebo capsules to be administered once a day for a total of 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — 5mg rapid release melatonin capsule
  Arms: Melatonin
Other: Placebo — matching placebo capsule
  Arms: Placebo

SUMMARY:
This is an 8-week randomized, double-blind, placebo-controlled, parallel, fixed-dose pilot clinical trial to test the effectiveness of melatonin treatment versus placebo on symptoms of Night Eating Syndrome (NES). The investigators will also look at the effect of melatonin treatment on weight, metabolic parameters and sleep parameters in individuals with NES.

DETAILED DESCRIPTION:
Night Eating Syndrome (NES) is a unique disorder characterized by a delayed pattern of food intake in which recurrent episodes of food consumption occurs after the evening meal and/or during nocturnal awakenings. Diagnostic criteria for NES include: (1) recurrent episodes of night eating, as manifested by eating after awakening from sleep or by excessive food consumption following the evening meal, (2) awareness of those eating episodes, and (3) significant distress or impairment caused by the disorder. Exclusion criteria are binge-eating disorder or another mental disorder, as well as medical disorders or medications that might better explain the disordered eating pattern. NES is also more common among patients with insomnia, eating disorders, and other psychiatric disorders. 100 participants with night eating syndrome will be recruited from the general population. They will be randomized to either a commercially available rapid-release formulation of melatonin (5 mg) or matching placebo capsules, that will be administered once a day for a total of 8 weeks. Participants will attend a screening appointment, a baseline assessment and additional research assessment visits every other week for the 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 65 years of age
2. English speaking
3. Meet DSM-V (Diagnostic and Statistical Manual - version 5) criteria for Night Eating Syndrome (NES)

Exclusion Criteria:

1. Unable to provide informed consent
2. Presence of alcohol/substance dependence
3. Presence of other eating disorders such as Binge Eating Disorder, Anorexia Nervosa.
4. Significant uncontrolled systemic illness (e.g. chronic renal failure, chronic liver disease, poorly controlled diabetes, poorly controlled congestive heart failure, chronic infectious disease, chronic autoimmune disease)
5. Women who are pregnant or breastfeeding
6. Allergy or hypersensitivity to melatonin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Change in Night Eating Syndrome Symptoms - Night Eating Symptom Scale (NESS) Total Score | 8 weeks
  Change in total score for the Night Eating Symptom Scale (NESS) from baseline to endpoint. Scores range from 0-52. Lower scores are better than higher scores.

SECONDARY OUTCOMES:
Change in body weight in kilograms during study duration. | 8 weeks
  Change in body weight in kilograms from baseline to endpoint.
Change in body mass index (BMI) during study duration | 8 weeks
  Change in body weight in kilograms from baseline to endpoint.
Change in waist circumference in centimeters during study duration. | 8 weeks
  Change in waist circumference in centimeters from baseline to endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data resulting from this award involving human subjects will be submitted to the NIMH Data Archive (NDA) - National Database for Clinical Trials Related to Mental Illness (NDCT) The Principal Investigator will work with NDA support staff to plan an appropriate data submission schedule and provide information on the steps for submission and sharing of data. Communication of this data sharing plan to appropriate research staff to ensure the timely submission of data. All human subject data provided will include an NDA Global Unique Identifier (GUID) and will not include personally identifiable information (PII). Analyzed data will be submitted no later than the time of publication. Even if a publication focuses on only part of an analyzed dataset, the entire analyzed dataset will be submitted when the first paper is published. All data made available for public use via NDA will be de-identified data.